CLINICAL TRIAL: NCT03277781
Title: Female Aneurysm Screening STudy
Acronym: FAST
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: 0573; 2016-001261-83 (EudraCT Number); PB-PG-0215-36027 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2017-08-29; First posted 2017-09-11 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2019-09

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Current smokers
  Interventions: Other: Screening
- Ex-smokers
  Interventions: Other: Screening
- Coronary heart disease
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Screening for AAA

SUMMARY:
An abdominal aortic aneurysm (AAA) is a swelling of the main blood vessel (aorta) in the abdomen. If the swelling gets too large the aorta can burst and this is usually fatal. In order to prevent rupture, AAA can be surgically repaired. This is usually carried out when the size of the AAA is more than 5.5cm in diameter as below this size, the risk of rupture is lower than the risk of surgery. AAA are usually asymptomatic before rupture but can easily and safely be diagnosed by ultrasound scanning. There is currently a national screening programme for men, but not women.

Women are not screened for AAA on the basis that the disease is less common in females. However, 33.6% of all deaths caused by ruptured AAA in England and Wales are in females (1109 female deaths)1. Death rates due to ruptured AAA in men have nearly halved over the last decade but the reduction in female deaths over the same time period is less than one third. Females with AAA are also 4-times more likely to rupture their aneurysm and have higher rates of complications and death after emergency surgery than men.

There are groups of females such as smokers, who are at high risk of AAA. The investigators have identified risk factors that are easily identifiable from general practice databases that may be able to identify women at high risk of AAA. In this research it will be determined whether it is feasible to select women for AAA screening using these risk factors, how many women in these high-risk groups attend if they are invited for AAA screening, and screen women to determine the numbers in the different risk groups who have AAA. This will allow the assessment of whether screening women for AAA could be clinically or cost effective and who would benefit the most. The investigators will also investigate if the siblings of patients with AAAs are at higher risk of disease by inviting them for screening too.

ELIGIBILITY:
Inclusion Criteria:

* As per group definitions

Exclusion Criteria:

* Any significant disease or disorder which, in the opinion of the Investigator or the patient's general practitioner, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Ages: 65 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: White women aged 65 to 74 with a history of smoking and/or coronary heart disease
Sampling Method: Non-Probability Sample
Enrollment: 5612 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Attendance | Day 1
  Proportion of women attending for AAA screening
Prevalence | Day 1
  Proportion of women who attend for screening who have an AAA

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No